CLINICAL TRIAL: NCT04143178
Title: Effectiveness of a Psychological Intervention Focused on Expressive Writing in Patients Undergoing to Kidney Transplant
Brief Title: Expressive Writing in Kidney Transplant Patients
Acronym: EWKTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Carlo Lai, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08/2019
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Kidney Transplant Rejection
Keywords: Expressive writing; Kidney transplant; Adherence; Alexithymia; Healthcare spending
MeSH Terms: conditions — Affective Symptoms

STUDY DESIGN:
Intervention Model Description: Five days after the transplant, to the expressive writing group participants has been asked to write for 3 consecutive days, for 20 minutes a day, their deepest emotions, thoughts and concerns about the disease and the transplant. They wrote in a silent room that guaranteed their privacy. The instructions followed the standard task of Pennebaker, creator of the technique (1986), translated and adapted for the specific hospital situation already proposed in a study on urological patients by Solano et al, 2007.
  Similarly, five days after the transplant, to the control group participants has been asked to write for 3 consecutive days 20 minutes a day on an assigned neutral theme (eg. describe 1 object in the room) as objectively as possible, without mentioning their emotions or thoughts related to it.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expressive Writing Group (Experimental): Writing group participants has been asked to write for 3 consecutive days, 20 minutes each days, all the deepest emotions and feelings related to the disease, the transplant, and their best expectations after the operation.
  Interventions: Other: Expressive Writing
- Control Group (Other): The control group participant has been asked to describe an objects in their room, in a neutral way, without mentioning emotions or feelings,for 3 consecutive days, 20 minutes each day.
  Interventions: Other: Neutral Writing

INTERVENTIONS:
Other: Expressive Writing — The expressive writing is a form of writing therapy developed primarily by James W. Pennebaker in the late 1980s consisting of writing about stressful and traumatic experience for 15-20 min for 3 consecutive days, including one's thoughts and feelings. The expressive writing allows people to express and process emotions, feelings, and thoughts related to the life events and consequent changes and this may favor a mental reorganization of the negative events, a greater expression and regulation of the emotions related to them. This intervention could provoke social, emotional, and consequently, psychophysical changes as is showed in patients with chronic diseases and cancer. In the present study, to all participants in the writing group, 5 days after the transplant, has been asked to write for 3 consecutive days, 20 minutes each days about their deepest emotions and feelings related to the chronic failure, the transplant and their expectations after that.
  Arms: Expressive Writing Group
Other: Neutral Writing — Five days after the transplant, to the control group participants has been asked to write for 3 consecutive days 20 minutes a day on an assigned neutral theme (eg. describe 1 object in the room) as objectively as possible, without mentioning their emotions or thoughts related to it.
  Arms: Control Group

SUMMARY:
Kidney transplantation is a replacement treatment for chronic renal failure that improves quality of life. However, it can be experienced as traumatic in relation to the changes it entails in terms of lifestyle, redefinition of one's body and social and family role. A negative personal experience could affect adherence to the treatment, a protective factor in reducing the risk of organ rejection and mortality. Some studies have shown the effectiveness of expressive writing in reducing the symptoms and management of the disease in patients undergoing surgery or suffering from cancer. It is hypothesized that this technique allows the processing of traumatic events linked to the disease, favoring an improvement in the expression and emotional regulation skills.

The aim of the present study was to evaluate the effectiveness of a psychological intervention focused on expressive writing on the post-operative course in patients underwent to kidney transplantation. Thirty-five patients were recruited at the kidney transplant center of the Policlinico Umberto I, Rome. The sample was divided into 2 groups: the psychological intervention focused on expressive writing group and the control group which carried out a neutral writing task. Each patient filled some self-report questionnaires and carried out blood analysis, before the operation, the day of discharge and at 3 month follow-up. The psychological intervention group was expected to have a greater improvement in the emotional skills, adherence and renal function, and a lower level of healthcare costs compared to the control group.

DETAILED DESCRIPTION:
Kidney transplantation is a replacement therapy in chronic renal failure which could allow a better quality of life. However, renal transplantation also represents an emotionally strong experience, which is associated with feelings of acceptance of the transplanted organ, change in lifestyle, side effects of pharmacotherapies, anxiety, depression, redefinition of one's body, as well as one's own social and family role. For these reasons it can be experienced as a traumatic event and be associated with an unfavorable post-operative course, in particular with regard to adherence to medical prescriptions and the consequent increase in the possibility of rejection.

Adherence, in fact, implies the correct management of drugs and the constant and assiduous presence at pre-established check-ups at the transplant center, taking the required exams and promptly reporting any complications. In kidney transplant patients, adherence to immunosuppressive therapies becomes fundamental to reduce the risk of organ rejection or, in the most extreme cases, the risk of death. Several studies show the importance of adherence to post-operative course treatment in different types of transplant. Furthermore, it has been shown that poor levels of adherence, recognized as a risk factor for organ rejection, are associated with an increase in healthcare costs.

Young age, depression, anxiety and avoidant-type adaptation strategies (eg avoiding the stressful event) are some of the risk factors of non-adherence in kidney transplant patients. Also alexithymia (known as the inability to identify and describe emotions), the inability to regulate intense emotional states, and attachment style, are associated with poor levels of post-transplant adherence.

Possemato and collaborators (2010), showed the efficacy of an intervention that uses expressive writing in the reduction of post-traumatic stress symptoms in kidney transplant patients. This technique seems to be effective also in patients with chronic pathologies and cancer, in particular in the reduction of symptoms , in the management of disease and psychophysical symptoms in cancer patients. The ways in which this technique acts are not yet clear, however it is hypothesized that the externalization and processing of traumatic events linked to the disease may favor an improvement in the ability to express emotions, and the reduction of negative thoughts and feelings associated. These studies suggest that using the technique of expressive writing in kidney transplant patients would allow them to externalize and process emotions, feelings and thoughts related to illness, transplantation and consequent changes (constant controls and therapies, sudden life style change, drug therapies and its effects, physical modifications), and this can favor a mental reorganization of negative events, a greater expression and emotions regulation, and an improvement in the interpersonal skills with family members and medical staff. Furthermore, this could be associated with a greater ability to cope with the consequences and psychophysical changes following transplantation and encourage greater levels of adherence with effects on the risk of organ rejection and health costs.

The objective of the study was to verify the effects of the expressive writing, on the post-operative course, in term of organ rejection, psychological well-being, adherence and healthcare spending in patients undergoing kidney transplantation.

Thirty-five patients were recruited at the kidney transplant center of the Policlinico Umberto I, Sapienza University of Rome. Each participant completed an informed consent form. The sample was divided into two groups in a randomized way. Of the 35 patients, 3 were excluded for not completing the task, due to logistical problems and due to the hospital situation, 1 refuse to perform the writing task, and finally 3 dropped to T2 (3rd post-transplant month). Of the remaining 28, 2 had an acute rejection before starting the writing task. The final sample is n = 26.

The study had 3 phases:

1. Pre-operative phase (T0)

   The time of admission, just before the kidney transplant. In this phase to all participants were asked socio-demographic information and specific characteristics of the pathology in progress (eg.duration of dialysis treatment, date of transplantation, onset of disease). Then, they completed the following self-administered questionnaires:

   Beck Depression Inventory (BDI) for the evaluation of depression, State Trait Anxiety Inventory I and II (STAI Y1 - STAI Y2) for the evaluation of trait and state anxiety, Toronto Alexythymia Scale 20-item (TAS-20) for assessing the ability to identify and describe one's emotions, Interpersonal Reactivity index (IRI) for the evaluation of empathy and the Health Locus of Control for the evaluation of the patient's beliefs on his state of health and a questionnaire for the evaluation of healthcare costs, built ad hoc.

   To assess the level of adherence, each patient answered to the following question: "Have you ever forgotten to take drugs prescribed by your treatment plan? "with dichotomous answer yes / no. Finally, in order to assess the pre-transplant renal function values, such as Creatinine, CDK-EPI and azotemia were collected.
2. Writing Phase (WP) Five days after the operation, patients belonging to the experimental group, performed the writing task related to their deepest emotions, thoughts and concerns focused on the disease and the transplant itself, for 3 consecutive days, for 20 minutes a day. They performed the writing session in a closed and silent room, which guaranteed their privacy. The instructions were according to the standard delivery by Pennebaker, creator of the technique, translated and adapted for the specific hospital situation already proposed in a study on urological patients by Solano et al. (2007). Instead, the control group performed the neutral writing task, related to the description of an object in their room, without mentioning emotions, but just describing in a neutral way what they saw, for 3 consecutive days, 20 minutes each day.
3. The day of discharge Phase (T1) and 4) three months follow up (T2) All participants filled the questionnaire completed before the operation and they had the blood analysis according to the hospital protocol for transplanted patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) of Italian nationality with sufficient level of education in order to understand the questionnaires and to carry out the writing task required by the protocol.

Exclusion Criteria:

* Patients with major psychopathology and/or cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Renal Function | 3 months
  In order to test the transplanted organ function the creatinine, CDK-EPI and azotemia level were measured through blood analysis at T0,T1,T2.
Alexithymia - difficulties in identifying, recognizing and describing emotions | 3 months
  In order to evaluate the level of alexithymia the TAS-20 was administered before the operation, the day of the discharge and 3 months after the transplant. It is a self-administered questionnaire, consisting of 20 items. The scale ranges between 20 to 100 and it allows to identify alexithymic (> 60), not alexithymic (< 51) and probably alexithymic patients (51-60).We expect that those patients undergoing expressive writing would have a lower score (<51) compared to control group patients.
Adherence | 3 months
  In order to assess the level of adherence, each patient had to answer to the following question: "Have you ever forgotten to take the drugs prescribed by your treatment plan?" with dichotomous answer yes / no
Healthcare spending | 3 months
  In order to test the healthcare spending to all participants were asked (through a specific questionnaire built ad hoc for the specific situation) the number of medical visits, the number of hospitalizations, the number of admissions to emergency room for acute episodes, the number of hospitalizations stay days in the last year, after the operation and 3 months later. The study hypothesized an lower number of medical visits, hospitalization's days and admissions to emergency room for those patients who performed the expressive writing task.

SECONDARY OUTCOMES:
Depressive symptoms | 3 months
  In order to test any variation in depressive symptoms the BDI -II was administered at T0,T1, and T2. The Scores 0-13 indicate an absence of depressive content, the scores between 14-19 a mild depression, the scores 27-29 a moderate grade depression and the scores 30-63: a severe depression. We expected a lover level of depression in all sample, and in particular lower level (0-13) in those who performed the expressive writing task.
Anxiety | 3 months
  In order to test any variation in anxiety level all participants completed STAI Y1, Y2 at T0, T1,T2. The scores between 80-71 represent very high level of state and trait anxiety, 70-51 represent medium-high level, 50-31 represent medium-low level and 30-20 none or very low level. We expected lower level of anxiety in all sample, but in particular lower level in those who performed the expressive writing task.
Empathy | 3 months
  In order to test the level of empathy the IRI questionnaire was administered at T0,T1,T2. It is a multidimensional scale composed of 28 self-report items designed to measure both cognitive and emotional components of empathy. The subscale scores range from 0 to 28. We expected higher level of empathy in those who performed the expressive writing task.
Resilience | 3 months
  In order to test the level of resilience, the CD-RISC Connor Davidson Resilience Scale was administered at T0,T1,T2. It is a self- administered questionnaire composed of 25 item and 5 subscales, with higher scores reflecting greater resilience. The score range from 0 to 100. We expected higher level of resilience in those who performed the expressive writing task.
Health Locus of control (HLC) | 3 months
  In order to test the patient's beliefs about the state of health, the Health Locus of Control test was administered at T0,T1,T2. It is a self- administered questionnaire composed of 11 item and 2 subscales (external locus of control and internal locus of control). The score ranges from 0 to 55. We expected higher level of internal locus of control in those who performed the expressive writing task.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Lai, Professor, Principal Investigator — Sapienza University of Rome, Italy
Locations (1):
- Azienda Policlinico Umberto I Sapienza University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data were collected in an excel database on the department of Dynamic and Clinical psychology laptop, protected by a password. The data are accessibile only to the Chief Investigator, the PhD student and the sub-investigator. The study protocol will be shared to other sub investigators involved in the study, but non the sensitive datas. The study report will be shared and published in a scientific journal, but the privacy of each participant will be respected according to the ethical committee established agreements.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 24 months
Access Criteria: The sensitive data are collected in an excel database on the department of Dynamic and Clinical psychology laptop, protected by a password. Each participant is identified by a personal numerical code, to guarantee them their privacy. All the sensitive data will be accessible only by the Chief investigator, the PhD student and the sub-investigator co-responsible of the study.

REFERENCES:
- [Background] De Pasquale C, Veroux M, Indelicato L, Sinagra N, Giaquinta A, Fornaro M, Veroux P, Pistorio ML. Psychopathological aspects of kidney transplantation: Efficacy of a multidisciplinary team. World J Transplant. 2014 Dec 24;4(4):267-75. doi: 10.5500/wjt.v4.i4.267. PMID 25540735
- [Background] Calia R, Lai C, Aceto P, Luciani M, Romagnoli J, Lai S, Gargiulo A, Citterio F. Effects of switching from twice-daily to once-daily tacrolimus formulation on quality of life, anxiety, and transplant benefit perception after kidney transplantation. Transplant Proc. 2011 May;43(4):1020-3. doi: 10.1016/j.transproceed.2011.03.048. PMID 21620041
- [Background] Calia R, Lai C, Aceto P, Luciani M, Camardese G, Lai S, Fantozzi C, Pietroni V, Salerno MP, Spagnoletti G, Pedroso JA, Romagnoli J, Citterio F. Emotional self-efficacy and alexithymia may affect compliance, renal function and quality of life in kidney transplant recipients: results from a preliminary cross-sectional study. Physiol Behav. 2015 Apr 1;142:152-4. doi: 10.1016/j.physbeh.2015.02.018. Epub 2015 Feb 11. PMID 25680476
- [Background] Gallo I, Garrino L, Di Monte V. [The use of expressive writing in the course of care for cancer patients to reduce emotional distress: analysis of the literature]. Prof Inferm. 2015 Jan-Mar;68(1):29-36. doi: 10.7429/pi.2015.681029. Italian. PMID 25837613
- [Background] Klein K, Boals A. Expressive writing can increase working memory capacity. J Exp Psychol Gen. 2001 Sep;130(3):520-33. doi: 10.1037//0096-3445.130.3.520. PMID 11561925
- [Background] Lai C, Aceto P, Luciani M, Fazzari E, Cesari V, Luciano S, Fortini A, Berloco D, Canulla F, Bruzzese V, Lai S. Emotional management and biological markers of dietetic regimen in chronic kidney disease patients. Ren Fail. 2017 Nov;39(1):173-178. doi: 10.1080/0886022X.2016.1256312. Epub 2016 Nov 15. PMID 27846784
- [Background] Buda B. Stephen J. Lepore & Joshua M. Smyth (Eds.) (2002). The Writing Cure: How Expressive Writing Promotes Health and Emotional Well-Being. By Bela Buda. Crisis. 2002 May;23(3):139. doi: 10.1027//0227-5910.23.3.139a. No abstract available. PMID 26200669
- [Background] Fallon M, Gould D, Wainwright SP. Stress and quality of life in the renal transplant patient: a preliminary investigation. J Adv Nurs. 1997 Mar;25(3):562-70. doi: 10.1046/j.1365-2648.1997.1997025562.x. PMID 9080284
- [Background] McGuire KM, Greenberg MA, Gevirtz R. Autonomic effects of expressive writing in individuals with elevated blood pressure. J Health Psychol. 2005 Mar;10(2):197-209. doi: 10.1177/1359105305049767. PMID 15723890
- [Background] Gremigni P, Bacchi F, Turrini C, Cappelli G, Albertazzi A, Bitti PE. Psychological factors associated with medication adherence following renal transplantation. Clin Transplant. 2007 Nov-Dec;21(6):710-5. doi: 10.1111/j.1399-0012.2007.00727.x. PMID 17988263
- [Background] Norman SA, Lumley MA, Dooley JA, Diamond MP. For whom does it work? Moderators of the effects of written emotional disclosure in a randomized trial among women with chronic pelvic pain. Psychosom Med. 2004 Mar-Apr;66(2):174-83. doi: 10.1097/01.psy.0000116979.77753.74. PMID 15039501
- [Background] Pabst S, Bertram A, Zimmermann T, Schiffer M, de Zwaan M. Physician reported adherence to immunosuppressants in renal transplant patients: Prevalence, agreement, and correlates. J Psychosom Res. 2015 Nov;79(5):364-71. doi: 10.1016/j.jpsychores.2015.09.001. Epub 2015 Sep 18. PMID 26526310
- [Background] Pennebaker JW, Beall SK. Confronting a traumatic event: toward an understanding of inhibition and disease. J Abnorm Psychol. 1986 Aug;95(3):274-81. doi: 10.1037//0021-843x.95.3.274. No abstract available. PMID 3745650
- [Background] Pisanti R, Lombardo C, Luszczynska A, Poli L, Bennardi L, Giordanengo L, Berloco PB, Violani C. Appraisal of transplant-related stressors, coping strategies, and psychosocial adjustment following kidney transplantation. Stress Health. 2017 Oct;33(4):437-447. doi: 10.1002/smi.2727. Epub 2016 Nov 9. PMID 27862894
- [Background] Prihodova L, Nagyova I, Rosenberger J, Majernikova M, Roland R, Groothoff JW, van Dijk JP. Adherence in patients in the first year after kidney transplantation and its impact on graft loss and mortality: a cross-sectional and prospective study. J Adv Nurs. 2014 Dec;70(12):2871-83. doi: 10.1111/jan.12447. Epub 2014 May 22. PMID 24853863
- [Background] Rebafka A. Medication Adherence After Renal Transplantation-a Review of the Literature. J Ren Care. 2016 Dec;42(4):239-256. doi: 10.1111/jorc.12181. Epub 2016 Sep 15. PMID 27629770
- [Background] Calia R, Lai C, Aceto P, Luciani M, Camardese G, Lai S, Amato G, Pietroni V, Salerno MP, Pedroso JA, Romagnoli J, Citterio F. Attachment style predict compliance, quality of life and renal function in adult patients after kidney transplant: preliminary results. Ren Fail. 2015 May;37(4):678-80. doi: 10.3109/0886022X.2015.1010989. Epub 2015 Feb 17. PMID 25687387
- [Background] Smyth JM, Stone AA, Hurewitz A, Kaell A. Effects of writing about stressful experiences on symptom reduction in patients with asthma or rheumatoid arthritis: a randomized trial. JAMA. 1999 Apr 14;281(14):1304-9. doi: 10.1001/jama.281.14.1304. PMID 10208146
- [Background] Solano L, Pepe L, Donati V, Persichetti S, Laudani G, Colaci A. Differential health effects of written processing of the experience of a surgical operation in high- and low-risk conditions. J Clin Psychol. 2007 Apr;63(4):357-69. doi: 10.1002/jclp.20355. PMID 17279528

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT04143178/Prot_SAP_000.pdf